CLINICAL TRIAL: NCT02602665
Title: Central Line Placement Study -EVALUATION OF LINE DEPTH AS A FACTOR IN NEED FOR LINE REPLACEMENT SECONDARY TO MALPOSITION
Brief Title: Central Line Placement-EVALUATION OF LINE DEPTH AS A FACTOR IN NEED FOR LINE REPLACEMENT SECONDARY TO MALPOSITION
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Design was not feasible
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Marcus Jarboe, Assistant Professor of Surgery and Assistant Professor of Radiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 98248
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Vascular Access Complication
Keywords: catheter placement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shallow catheter tip placement (Experimental): Patients randomized to shallow tip placement will have the tip of the catheter placed approximately one vertebral body above to even with the carina.
  Interventions: Procedure: Shallow catheter tip placement
- Deep catheter tip placement (Experimental): Patients randomized to deep tip placement will have the tip of the catheter placed 1.5 to 2.5 vertebral bodies below the carina.
  Interventions: Procedure: Deep catheter tip placement

INTERVENTIONS:
Procedure: Shallow catheter tip placement — for shallow placement tip of catheter placed 1 vertebral body above to even with the carina
  Arms: Shallow catheter tip placement
Procedure: Deep catheter tip placement — deep placement catheter tip is placed 1.5 to 2.5 vertebral bodies below the carina
  Arms: Deep catheter tip placement

SUMMARY:
This is a single center, randomized, controlled trial in which tunneled central line catheters will be placed in two distinct, select positions. The catheter tip position will then be followed up prospectively after placement to determine whether there is any malpositioning of the tip and if one placement is better than the other.

DETAILED DESCRIPTION:
Optimal central line placement is vital to catheter longevity. If malpositioned, the catheter may need to get replaced, potentially causing additional morbidity to the patient and additional cost to the healthcare system. In our department, a retrospective study looking at catheter tip position at inital placement and incidence of malposition. In this study, 404 catheter placements were reviewed, and a total of 162 (40.1%) were replaced. Out of the 162 replaced, 36 (22.2%) were replaced secondary to malposition. From this study, we were also able to conclude that catheter tips placed in a deeper position, approximately one and a half vertebral bodies below the carina, were less likely to be malpositioned in the future upon radiographic review.

Current standard of care does not dictate positioning of the line in a specific loacation. In the presence of these findings, we are proposing to conduct a single center randomized control trial in which tunneled central line catheters will be placed in two distinct, select positions. After informed consent is obtained from the patient and family, they will be randomized to one of two treatment groups. The shallow group will have the tip of the catheter located approximately one vertebral body above the carina. The deep group will have the catheter tip placed 1.5 to 2.5 vertebral bodies below the carina. Central line placement will be performed under fluoroscopy in the operating room to optimize catheter placement. Chest X ray in the post operative area will be used to confirm catheter tip position. The catheter tip position will then be followed up prospectively using chest X ray films at or within three months after placement to determine whether there is any malpositioning of the tip.

ELIGIBILITY:
Inclusion Criteria:

* Children from 0-18 years of age needing a tunneled central line (port or broviac) for treatment of their disease.

Exclusion Criteria:

* Wire exchanged lines
* Non ultrasound placed lines, femoral lines, saphenous vein lines, and cut downs
* Short gut syndrome children < 1 year of age

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-28 (Estimated); Study Completion 2021-12-28 (Estimated)

PRIMARY OUTCOMES:
Malposition | 90 days
  The primary outcome measure of this study is to determine whether the position of the tip during central line placement plays a role in malposition during further evaluation of these patients. This will be determined with chest X-ray done at or within 90 days after line insertion. All non-ultrasound guided lines and those placed by cut down procedure will be tallied in a prospective manner to calculate the number of lines placed without radiological guidance. Number of attempts required to place the line (number of times the needle is removed exterior to the skin, i.e. number of skin punctures.)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Jarboe, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No